CLINICAL TRIAL: NCT03444025
Title: Prospective Phase II Randomized Trial of Evaluating the Effect of Adding LHRH Analogue to the Neoadjuvant Chemotherapy Treatment of Triple Negative Breast Cancer on Pathologic Complete Response (pCR) Rates
Brief Title: Neoadjuvant Goserelin for Triple Negative Breast Cancer
Acronym: NeoGONT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Kyrillus S Shohdy, Dr., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-11
Record Dates: First submitted 2018-02-18; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer Triple Negative
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Goserelin 3.6 mg depot injection will be administered subcutaneously every month along with standard chemotherapy regimen: AC-P: Doxorubicin 60 mg/m2 IV plus cyclophosphamide 600 mg/m2 every 3 weeks for four cycles, followed by paclitaxel 80 mg/m2 by 1 hour infusion every week for 12 weeks. Each cycle is 21 days.
  Interventions: Drug: Goserelin
- Group B (No Intervention): Standard chemotherapy regimen: AC-P: Doxorubicin 60 mg/m2 IV plus cyclophosphamide 600 mg/m2 every 3 weeks for four cycles, followed by paclitaxel 80 mg/m2 by 1 hour infusion every week for 12 weeks. Each cycle is 21 days.

INTERVENTIONS:
Drug: Goserelin — Goserelin is Luteinizing hormone releasing hormone (LHRH) analogue.
  Other Names: Zoladex
  Arms: Group A

SUMMARY:
This is a phase II randomized trial that will evaluate the effect of adding LHRH analogue, goserelin, to the standard neoadjuvant chemotherapy to patients with triple negative breast cancer. Targeting LHRH might decrease resistance to chemotherapeutic agents in the neoadjuvant setting and increases clinical and pathological response rates. Additionally, exploring potential surrogate markers (as AR and LHRH receptors) for molecular distinct subtypes of TNBC.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy (NACT) is the mainstay of treatment of locally advanced TNBC and some selected early cases followed by surgery with or without adjuvant radiotherapy. NACT is aimed to induce pathologic complete response (pCR) in tumor and lymph nodes, pCR is proofed to be a surrogate and reliable predictive factor of survival rates in TNBC. This study will evaluate the effect of adding LHRH analogue, goserelin, to the standard neoadjuvant chemotherapy. Following completion of neoadjuvant therapy, patients will undergo breast conservative surgery or mastectomy. Post-neoadjuvant chemotherapy axillary staging will be required, but the choice of the procedure will be at the physician's discretion. Postoperative radiation therapy will be given at the physician's discretion. The use of partial breast irradiation techniques will not be allowed. The primary endpoint will be the rate of pathologic complete response. The secondary endpoints will be 3-year-disease free survival, clinical response and toxicity. Exploratory endpoints will be correlation of the LHRH receptor expression level with the pCR. The sample size for the trial will be 180 patients accrued over a period of 2 years. Definitive analysis of the primary endpoints is expected at year 3.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women between 18 and 60 years.
2. Histologically proven, newly diagnosed invasive carcinoma of breast.
3. Tumors must be ER, PgR negative and HER2-neu negative.
4. Stage II or III breast cancer that is indicated for neoadjuvant systemic chemotherapy.

Exclusion Criteria:

1. pregnant females at time of diagnosis of breast cancer.
2. bilateral breast cancer.
3. already received treatment for breast cancer including surgery, radiation, cytotoxic, or endocrine therapy
4. history or concomitant diagnosis of another primary malignancy.
5. concurrent treatment with oral contraceptives or hormone replacement therapy (OCPs or HRT must be stopped at least 4 weeks prior to randomization).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 180 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response rate | 6 months
  The primary endpoint will be the pathologic complete response rate (pCR), defined as no residual invasive tumor in both the breast and axilla (and including in situ residual; ypT0/is, ypN0).

SECONDARY OUTCOMES:
LHRH-positive and/or AR-positive Rate | 6 months
  Incidence of LHRH-positive and/or AR-positive cases among TNBC
Relapse-free Survival | 3 years
  Estimated 3 years RFS rates in the 2 arms (RFS events will include locoregional recurrence, distant recurrence, contralateral breast cancer and death from any cause).
Objective response rate | 6 months
  Clinical and radiological ORRs
Adverse events | 6 months
  All grade and high grade adverse events rate in both arms
Ovarian failure rate | 2 years
  Ovarian failure rates at 2 years in both groups (defined as the absence of menses in the preceding 6 months and levels of follicle-stimulating hormone (FSH) in the postmenopausal range).

IPD SHARING:
Plan to Share IPD: Undecided